CLINICAL TRIAL: NCT00351455
Title: Watchful Waiting of Incisional Hernias: A Prospective Trial
Brief Title: Watchful Waiting of Incisional Hernias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Daniel Musher, Distinguished Service Professor of Medicine, Baylor College of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H-18609
Record Dates: First submitted 2006-07-07; First posted 2006-07-12 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Incisional Hernia; Ventral Hernia; Umbilical Hernia
Keywords: hernia; incisional hernia; ventral hernia; umbilical hernia
MeSH Terms: conditions — Incisional Hernia; Hernia, Ventral; Hernia, Umbilical; Hernia | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: smoking cessation
Behavioral: tighter diabetic control
Behavioral: diet and exercise program

SUMMARY:
This study is being conducted to gain a better understanding of the quality of life for patients with a diagnosis of primary and recurrent incisional hernias and 1) who decline to have surgery to repair the hernia or 2) patients who cannot have surgery because their health will not allow them or 3O if surgery to repair the hernia is completed. A comparison will be made between those who receive surgery and those who do not.

DETAILED DESCRIPTION:
This study is being conducted to gain a better understanding of the quality of life for patients with a diagnosis of primary and recurrent incisional hernias and 1) who decline to have surgery to repair the hernia or 2) patients who cannot have surgery because their health will not allow them or 3O if surgery to repair the hernia is completed. A comparison will be made between those who receive surgery and those who do not.

Subjects will fill out three survey forms on quality of life and pain at baseline and again at six and 12 months. Measurements of change in hernia size will be made, life-style changes such as smoking cessation, weight-loss, tighter control of diabetes will be initiated for outcome comparison with controls.

ELIGIBILITY:
Inclusion Criteria:

1. abdominal hernia greater than 3 cm2
2. 18 years of age
3. able to give informed consent

Exclusion Criteria:

1. abdominal hernia less than 3 cm2 or greater than 127 cm2
2. unable to return to clinic for follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-05; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Develop guidelines for hernia repair

SECONDARY OUTCOMES:
To measure if life-style changes lower need for hernia repair

CONTACTS AND LOCATIONS:
Overall Officials: Charles Bellows, III, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States